CLINICAL TRIAL: NCT03405142
Title: A Phase II Study Evaluating Panitumumab-IRDye800 vs. Sentinel Node Biopsy and (Selective) Neck Dissection for Metastatic Lymph Node Identification in Patients With Head and Neck Cancer
Brief Title: Panitumumab-IRDye800 Compared to Sentinel Node Biopsy and (Selective) Neck Dissection in Identifying Metastatic Lymph Nodes in Patients With Head&Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eben Rosenthal (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Eben Rosenthal, Professor of Otolaryngology, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-43013; NCI-2017-02425 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ENT0065 (Other: OnCore Number); P30CA124435 (NIH); R01CA190306 (NIH)
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Results first posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Squamous Cell Carcinoma of the Head and Neck (SCCHN); Head and Neck Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- T1 or T2 stage and node-negative (Experimental): T1 or T2 stage primary tumor and node-negative (ie, cN0)
  Interventions: Drug: Panitumumab-IRDye800; Drug: Lymphoseek
- Any T stage and node-positive (Experimental): Any T stage tumor and node-positive (ie, cN+)
  Interventions: Drug: Panitumumab-IRDye800

INTERVENTIONS:
Drug: Panitumumab-IRDye800 — Intravenous (IV) panitumumab-IRDye800 (50 mg) 1 to 5 days prior to surgery (lymphadenectomy). Panitumumab dose is < 1/12 of the therapeutic dose.
  Other Names: Panitumumab IRDye 800; RDye800-Panitumumab Conjugate
Drug: Lymphoseek — Local, peri-tomoral injection with 2 mCi Lymphoseek (99mTc Tilmanocept) (as 4 x 0.1 mL injections of Lymphoseek solution
  Other Names: 99mTc-Diethylenetriamine Pentaacetic Acid-Mannosyl-Dextran; 99mTc-DTPA-Mannosyl-Dextran; Technetium Tc 99m-labeled Tilmanocept
  Arms: T1 or T2 stage and node-negative

SUMMARY:
This phase 2 trial studies how well panitumumab-IRDye800 works in identifying head and neck cancer that has spread to the lymph nodes in patients with head and neck cancer. Panitumumab-IRDye800 may help surgeons to identify metastatic lymph nodes during surgical removal of the primary tumor and/or lymph nodes of the neck with equal or better accuracy than the current methods.

DETAILED DESCRIPTION:
Detecting progression of squamous cell carcinoma of the head and neck (SCCHN) is clinically challenging, with the transition from Stage 2 (no metastasis) to Stage 3 or 4 (minimally to significantly metastatic) representing a significant and adverse clinical milestone. SCCHN often spreads by movement of metastatic cells through the lymphatic system. Often, these cells are retained in various lymph nodes (LNs), of which there are over 150 on each side of the head and neck. Logically, the objective of neck dissection would be the removal of obvious cancer and any LNs containing metastatic cells. However, with visual or even radiologic identification of cancerous LNs was challenging at best, definitive assessment of the spread of the cancer must be made on excised tissue in the clinical laboratory by pathologic assessment. Historically, a marker of successful neck dissection for SCCHN was excision of sufficient LNs such that the extent of tumor-positive LNs would be demonstrated by pathology. Accordingly, many LNs are excised that turn out to be negative for invasive tumor cells. Unfortunately, neck dissection is often accompanied by significant morbidity, such as shoulder dysfunction or injury to the cranial nerve XI or other nerves causing persistent pain, as well as anatomic deformities such as scapular flaring, droop, and protraction. In recent years, a more limited dissection procedure known as sentinel lymph node biopsy (SNB) has become common, with the advantage of being less invasive, and targeted to only the LNs believed to the primary drainage of the tumor. Sentinel lymph nodes are those believed to be most likely to collect tumor cells migrating from the tumor lesion. The goal of SNB is a more precise identification of those LNs that have or are likely to have metastatic cells, with fewer LNs collected and less morbidity. Pathological assessment of the SNBs enhances clinical decision making for further treatment. While SNB represents an overall improvement, there remains opportunity for better detection of metastatic LNs with less morbidity.

In this study, the specific medical imaging scan is known as lymphoscintigraphy and is conducted as single-photon emission computerized tomography (SPECT) scan with computed tomography (CT), collectively "SPECT/CT" using the radiolabel Lymphoseek (99mTc Tilmanocept). Lymphoseek is administered as 4 injections to LNs that are in the immediate vicinity of the known tumor lesion.

The surgical procedure is known as lymphadenectomy, meaning excision of lymph nodes. In this study, the excised lymph nodes are those suspected as being positive for malignancy and the basis of they as SPECT/CT lymphoscintigraphy.

The panitumumab-IRDye800 agent is intended to bind to cancer cells, and enable detection of those cells on the basis of IRDye800 fluorescence. The panitumumab-IRDye800 is administered as an intravenous infusion over 15 minutes. The label is specific to a marker on tumor cells, and migrates through the body and adheres to cancer cells, permitting their identification visually or by fluorescence detectors. Immediately before and after excision, the area around the lymph nodes are evaluated for the fluorescent signal of the panitumumab-IRDye800. Additional areas of panitumumab-IRDye800 may be excised. The potential advantage of panitumumab-IRDye800 labeling is that signaling is assessed intraoperatively, and this may enable more accurate and more precise determination of the tumor in LNs and other tissue.

In this study, participants with SCCHN that is T1 or T2 stage and node-negative (ie, cN0) (Cohort 1) will undergo labeling procedures with Lymphoseek (99mTc Tilmanocept), a regular medical care radiolabel and also investigational panitumumab-IRDye800. Participants whose SCCHN is node positive and any T stage (Cohort 2) can participate and undergo labeling with investigational panitumumab-IRDye800 alone.

PRIMARY OBJECTIVES:

To determine if near-infrared fluorescence imaging of panitumumab-IRDye800 can identify metastatic disease in regional neck lymph nodes of patients with head and neck squamous cell carcinoma (HNSCC).

SECONDARY OBJECTIVES:

Determine if panitumumab-IRDye800 can identify sentinel nodes with the same accuracy as technetium Tc 99m-labeled tilmanocept (Lymphoseek).

OUTLINE:

Beginning 2-5 days before surgery, patients receive panitumumab IRDye800 intravenously (IV) over 60 minutes. On the day before surgery, patients also receive technetium Tc 99m-labeled tilmanocept via injection and undergo lymphoscintigraphy and single photon emission computed tomography/computed tomography (SPECT/CT).

After completion of study, patients are followed up for 30 days.

ELIGIBILITY:
INCLUSION CRITERIA:

* Biopsy-confirmed diagnosis of squamous cell carcinoma of the head and neck
* Patients with recurrent disease or a new primary will be allowed
* Planned standard of care surgery with curative intent for squamous cell carcinoma

  * Cohort 1: T1-T2 stage tumor diagnosis, any subsite within the head and neck that is amenable to local sentinel node tracer injection, and scheduled to undergo surgical resection of the tumor, including a sentinel node biopsy
  * Cohort 2 (neck dissection only): Diagnosis with any T-stage, any subsite within the head and neck that are scheduled to undergo surgical resection, including a (modified) neck dissection
* Age ≥ 19 years
* Karnofsky performance status of at least 70% or ECOG/Zubrod level 1
* Have acceptable hematologic status, coagulation status, kidney function, and liver function including the following clinical results:
* Hemoglobin ≥ 9 gm/dL
* White blood cell count > 3000/mm³
* Platelet count ≥ 100,000/mm³
* Serum creatinine ≤ 1.5 times upper reference range

EXCLUSION CRITERIA:

* Received an investigational drug within 30 days prior to first dose of panitumumab-IRDye800
* Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); significant liver disease; or unstable angina within 6 months prior to enrollment
* History of infusion reactions monoclonal antibody therapies
* Pregnant or breastfeeding
* Magnesium or potassium lower than the normal institutional values
* Receiving class IA (quinidine, procainamide) or class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents
* History or evidence of interstitial pneumonitis or pulmonary fibrosis
* Hypersensitivity to dextran and/or modified forms

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2021-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred M Baik, Principal Investigator — Stanford Cancer Institute Palo Alto
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T1 or T2 Stage and Node-negative | Any T Stage and Node-positive
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T1 or T2 Stage and Node-negative | Any T Stage and Node-positive | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 2 | 0 | 2
Age, Continuous [Median (Full Range); unit: years] | 76.5 [71.5 to 81.5] | 61.6 [61.6 to 61.6] | 71.5 [61.6 to 81.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Detection of Malignancy in Excised Lymph Nodes by Pathology or Labeling With Lymphoseek and/or Panitumumab-IRDye800
Description: After administration of panitumumab-IRDye800 alone or with Lymphoseek, lymph nodes potentially containing malignant tumor cells were surgically removed, and the lymph node tissue was evaluated for panitumumab-IRDye800 fluorescence intensity. For each subject, the 5 lymph nodes with the strongest fluorescence signal were tabulated against the Lymphoseek and histopathologic findings for those specific lymph nodes. For each of the 3 modalities, a positive finding is considered indicative of malignancy. The outcome is reported as the number of positive findings by modality for each cohort. The outcome is a number without dispersion.
Time Frame: Up to 30 days
Measure: Number; unit: Lymph nodes
Units Other Than Participants: Lymph nodes
Arm/Group | T1 or T2 Stage and Node-negative | Any T Stage and Node-positive
Number analyzed (Participants) | 2 | 1
Number analyzed (Lymph nodes) | 10 | 5
Lymph nodes
  Panitumumab-IRDye800 | 10 | 5
  Lymphoseek | 3 | NA — Lymphoseek not administered to this cohort.
  Histopathology | 2 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | T1 or T2 Stage and Node-negative | Any T Stage and Node-positive
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT03405142/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/42/NCT03405142/ICF_001.pdf